CLINICAL TRIAL: NCT00988403
Title: Investigation of Dietary Absorptive Capacity of Fructans in Healthy Subjects - A Randomized, Double-Blind Dose Response Study
Brief Title: Investigation of Dietary Absorptive Capacity of Fructans in Healthy Subjects - A Dose Response Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: American Gastroenterological Association Foundation (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Fructan
Record Dates: First submitted 2009-09-22; First posted 2009-10-02 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fructan - 7.5 (Experimental): Subjects will consume 7.5 grams of fructan
  Interventions: Dietary Supplement: Fructan - 7.5
- Fructan - 10 grams (Experimental): Subjects will consume 10 grams of fructan
  Interventions: Dietary Supplement: Fructan - 10
- Fructan - 12.5 grams (Experimental): Subjects will consume 12.5 grams of fructan
  Interventions: Dietary Supplement: Fructan - 12.5
- 5 grams Fructan (Experimental): Experimental - 5 grams Fructan
  Subjects will consume 5 grams of Fructan.
  Interventions: Dietary Supplement: Fructan -- 5 grams

INTERVENTIONS:
Dietary Supplement: Fructan - 7.5 — Subjects will consume 7.5 grams of fructan
  Other Names: 7.5 grams of Inulin
  Arms: Fructan - 7.5
Dietary Supplement: Fructan - 10 — Subjects will consume 10 grams of fructan
  Other Names: 10 grams of Inulin
  Arms: Fructan - 10 grams
Dietary Supplement: Fructan - 12.5 — Subjects will consume 12.5 grams of fructan
  Other Names: 12.5 grams of Inulin
  Arms: Fructan - 12.5 grams
Dietary Supplement: Fructan -- 5 grams — Subjects will consume 5 grams fructan.
  Other Names: 5 grams of Inulin
  Arms: 5 grams Fructan

SUMMARY:
Fructan is a carbohydrate polymer that is composed of fructose and a terminal glucose moiety . Fructans are naturally found in artichokes (6.1 grams/serving), leeks (5.9 grams/serving), onion bulbs (1.01 grams/serving), flour (4.0 grams/serving), garlic (.52 grams/serving), watermelon (.92 grams/serving), nectarines (.27 grams/serving) and white peaches (.50 grams/serving). Because fructans are present in many common foods, people typically ingest high levels of fructan. The most common structural forms of fructan are inulin, levanare and geraminan . The human body absorbs only 5% of fructan, however it is estimated that the daily intake in the USA may vary between 1-20 grams, and possibly higher due to the recently discovered benefits of inulins . Dietary trends indicate that high levels of fructans are common in the European and American diet, as more wheat based products such as breakfast cereal, pasta, and bread are consumed.

Fructans may not be well tolerated by some subjects and its malabsorption may result in gastrointestinal (GI) symptoms such as heartburn, belching, abdominal pain, diarrhea, gas, and bloating; and this is especially true when higher doses are ingested. Unlike glucose, fructans are not efficiently digested or absorbed by the small intestine. The mechanism for malabsorption is related to the inability to hydrolyze glycosidic linkages in the complex polysaccharide, resulting in the delivery of malabsorbed fructans to the large bowel1. In the colon, the malabsorbed fructans are rapidly fermented, and byproducts of this fermentation include H2, CH4, and other gases that may contribute to bowel symptoms. Furthermore, the small molecular nature of fructans results in an osmotic effect which draws more water into the small intestine and causes bloating and diarrhea.

Ingestion of high doses of fructans can cause symptoms in healthy adults, but may cause more bothersome symptoms in subjects with Irritable Bowel Syndrome (IBS). Earlier studies have identified that IBS affects between 10 and 15% of the population in the United States. Ingestion of 10-20 grams of fructan daily may cause symptoms of IBS, and restricting fructan intake in a diet may reduce symptoms in a variety of gastrointestinal disorders. One study recently published found that dietary restriction of fructan and fructose was responsible for symptomatic improvement in patients with IBS.

Hypothesis:

The investigators hypothesize that healthy individuals will absorb fructan 7.5 gram and 10 gram doses, and will experience malabsorption at the 12.5 gram fructan dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between the ages of 18-70 years, with no previous history of gastrointestinal problems or any other ailments, no history of gastrointestinal surgery except appendectomy, cholecystectomy, caesarean section, hysterectomy and currently not using any medication except contraceptive pill, multivitamin, or aspirin.
* They will be asked to fill out a Review of Systems health history (Appendix 2) and the Mayo Clinic Bowel Disease Questionnaire (Appendix 3) and will undergo a routine physical examination. Only patients who are asymptomatic and deemed healthy from the aforementioned screening procedure will be eligible.

Exclusion Criteria:

* Currently taking medication for any ailment including OTC medication (excluding aspirin, multivitamins, and oral contraceptives)
* History of gastrointestinal problems including bloating, gas, food intolerances or reflux symptoms
* Any major abdominal surgery (except appendectomy, cholecystectomy, caesarean section, hysterectomy) or coexisting medical problem
* Known food allergies
* Prisoners
* Cognitive Impairment or any other inability to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2011-08-31 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Hydrogen and Methane Concentration levels | 3 visits over a 1 month period
  Measure breath sample concentration for hydrogen and methane levels in parts per million

SECONDARY OUTCOMES:
Production of GI Symptoms | 3 visits over a 1 month period
  Production of bothersome GI symptoms such as gas, bloating, cramping or abdominal pain during breath test. Symptoms were mesured using a validated symptom questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Satish Rao, MD, PhD, Principal Investigator — Augusta University
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States